CLINICAL TRIAL: NCT00701519
Title: The Prevalence of Sleep Disordered Breathing in Hospitalized Patients With Acutely Decompensated Heart Failure Syndrome
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Rami Khayat, Associate Professor-Clinical, Ohio State University
Other Study IDs: 2007H0055
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Sleep Apnea; Congestive Heart Failure; Heart Failure
Keywords: CHF,; Sleep apnea,; Obstructive sleep apnea,; Heart failure
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
OSA is associated with large negative swings in the intrathoracic pressure, significant increase in the sympathetic nerve activity and repetitive surges in blood pressure, along with episodic hypoxia and hypercapnea (8,9). These autonomic and respiratory changes may increase the cardiac muscle workload, cardiac dysrrhythmia, and exacerbate ischemia (10,11,12). Treatment with CPAP is the most successful therapeutic modality available for OSA. It is still not clear whether establishing the diagnosis of OSA and initiating treatment with CPAP while still in the hospital carries any benefit in the management of patients with acute heart failure. This study will evaluate the effect of work up and treatment of OSA on the outcome of patients hospitalized with acute CHF.

DETAILED DESCRIPTION:
Congestive heart failure affects 2.3% of the population (approximately 4,900,000) with an incidence of 10 per 1,000 of the population after the age of 65 (1). The admission rate for patients with heart failure is on the rise, so is the mortality associated with it and its national annual bill, now exceeding $21 billion (1). Obstructive Sleep Apnea (OSA) is present in 11-37% of patients with heart failure (2,3), and tends to increase in severity when the heart failure is less controlled (4, 5). Therefore, the actual prevalence of OSA in patients hospitalized with acute heart failure is likely higher. There is now evidence that treatment of OSA with nasal Continuous Positive Pressure (nCPAP) in outpatients with stable heart failure improves left ventricular ejection fraction, and quality of life (6), and confers a reduction in fatal and non-fatal cardiovascular events (7). However, there has not been any evaluation of the role of diagnosis and treatment of OSA in patients hospitalized with acute heart failure. This uncertainty about the true prevalence and role of OSA in exacerbations of heart failure, and the role of its treatment in the acute setting may explain why aggressive diagnostic and therapeutic strategy for OSA in patients admitted to the hospital with acute heart failure is not part of the standard clinical practice in acute care centers. Given the rising admission rate, and mortality associated with heart failure, an evaluation of the role of OSA and its treatment in this patient population is highly significant.

The significance of this question resides mainly in the best approach to diagnosis and treatment of SDB in this high risk and vulnerable population. Should every patient wit heart failure undergo a polysomnography to diagnose a highly likely underlying SDB, and trigger appropriate treatment? The cost of polysomnography and the access to sleep laboratory makes it almost prohibitive to pursue such an approach. An approach that combines evaluation of risk factors and an abbreviated portable study may be adequate and certainly less expensive. Our OSU- Sleep Heart program was established to deliver expedient diagnosis and treatment of SDB to patients with heart failure. In the published literature, there are not adequate data to guide the delivery of Sleep services in this patient population. Our program aims at targeting every heart failure patient with validated questionnaires and screening ambulatory sleep studies. The sensitivity and specificity of such a surveillance approach will need to be evaluated against the reference standard, the polysomnography. Therefore this protocol aims to evaluate the negative and positive predictive value of our clinical program.

ELIGIBILITY:
Inclusion Criteria:

* OSU Heart Failure Patient
* Able to Complete Survey

Exclusion Criteria:

* Neurological Deficit
* No Heart failure
* Less than 18 yrs old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient with heart failure at the OSU is offered the opportunity to receive free screening for sleep apnea.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2007-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The risk and presence of sleep apnea in heart failure out patients. | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Rami N Khayat, MD, Principal Investigator — The Ohio Sate University
Locations (1):
- The Ohios State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1- Heart Disease and Stroke-Statistics, American Heart Association, 2005 update
- [Background] Javaheri S, Parker TJ, Liming JD, Corbett WS, Nishiyama H, Wexler L, Roselle GA. Sleep apnea in 81 ambulatory male patients with stable heart failure. Types and their prevalences, consequences, and presentations. Circulation. 1998 Jun 2;97(21):2154-9. doi: 10.1161/01.cir.97.21.2154. PMID 9626176
- [Background] Sin DD, Fitzgerald F, Parker JD, Newton G, Floras JS, Bradley TD. Risk factors for central and obstructive sleep apnea in 450 men and women with congestive heart failure. Am J Respir Crit Care Med. 1999 Oct;160(4):1101-6. doi: 10.1164/ajrccm.160.4.9903020. PMID 10508793
- [Background] Skinner MA, Choudhury MS, Homan SD, Cowan JO, Wilkins GT, Taylor DR. Accuracy of monitoring for sleep-related breathing disorders in the coronary care unit. Chest. 2005 Jan;127(1):66-71. doi: 10.1378/chest.127.1.66. PMID 15653964
- [Background] Solin P, Bergin P, Richardson M, Kaye DM, Walters EH, Naughton MT. Influence of pulmonary capillary wedge pressure on central apnea in heart failure. Circulation. 1999 Mar 30;99(12):1574-9. doi: 10.1161/01.cir.99.12.1574. PMID 10096933
- [Background] Mansfield DR, Gollogly NC, Kaye DM, Richardson M, Bergin P, Naughton MT. Controlled trial of continuous positive airway pressure in obstructive sleep apnea and heart failure. Am J Respir Crit Care Med. 2004 Feb 1;169(3):361-6. doi: 10.1164/rccm.200306-752OC. Epub 2003 Nov 3. PMID 14597482
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Katragadda S, Xie A, Puleo D, Skatrud JB, Morgan BJ. Neural mechanism of the pressor response to obstructive and nonobstructive apnea. J Appl Physiol (1985). 1997 Dec;83(6):2048-54. doi: 10.1152/jappl.1997.83.6.2048. PMID 9390980
- [Background] Morgan BJ, Denahan T, Ebert TJ. Neurocirculatory consequences of negative intrathoracic pressure vs. asphyxia during voluntary apnea. J Appl Physiol (1985). 1993 Jun;74(6):2969-75. doi: 10.1152/jappl.1993.74.6.2969. PMID 8365996
- [Background] Magder SA, Lichtenstein S, Adelman AG. Effect of negative pleural pressure on left ventricular hemodynamics. Am J Cardiol. 1983 Sep 1;52(5):588-93. doi: 10.1016/0002-9149(83)90032-2. PMID 6613883
- [Background] Stoohs R, Guilleminault C. Cardiovascular changes associated with obstructive sleep apnea syndrome. J Appl Physiol (1985). 1992 Feb;72(2):583-9. doi: 10.1152/jappl.1992.72.2.583. PMID 1559936
- [Background] Hanly P, Sasson Z, Zuberi N, Lunn K. ST-segment depression during sleep in obstructive sleep apnea. Am J Cardiol. 1993 Jun 1;71(15):1341-5. doi: 10.1016/0002-9149(93)90552-n. PMID 8498378
- [Background] Roebuck T, Solin P, Kaye DM, Bergin P, Bailey M, Naughton MT. Increased long-term mortality in heart failure due to sleep apnoea is not yet proven. Eur Respir J. 2004 May;23(5):735-40. doi: 10.1183/09031936.04.00060404. PMID 15176689